CLINICAL TRIAL: NCT02105714
Title: Diagnosis of Neglected Tropical Diseases (NTDs) in Patients Presenting With Persistent Digestive Disorders (≥2 Weeks) in Côte d'Ivoire, Indonesia, Mali and Nepal
Brief Title: Diagnosis of Neglected Tropical Diseases Among Patients With Persistent Digestive Disorders
Acronym: NIDIAGDigest
Status: Completed | Type: Observational
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other); B.P. Koirala Institute of Health Sciences (Other); Université Félix Houphouët-Boigny (Unknown); Institut de Recherche en Santé Publique, France (Other); Gadjah Mada University (Other)
Responsible Party: Sponsor
Other Study IDs: WP2-01-DIG
Record Dates: First submitted 2014-03-21; First posted 2014-04-07 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Soil-transmitted Helminthiasis; Schistosomiasis; Strongyloidiasis; Shigellosis; Intestinal Salmonellosis; Campylobacteriosis; Aeromonas Spp. Infections; Giardiasis; Amoebiasis; Dientamoebiasis; Cryptosporidium Spp. Infections
Keywords: Diarrhoea; Abdominal pain; Bacterial; Protozoal; Helminth
MeSH Terms: conditions — Schistosomiasis; Strongyloidiasis; Dysentery, Bacillary; Campylobacter Infections; Giardiasis; Amebiasis; Dientamoebiasis; Diarrhea; Abdominal Pain | interventions — Multiplex Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ethanol-preserved human stool specimens
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Stool culturing for pathogenic bacteria
Procedure: Kato-Katz technique
Procedure: Baermann technique
Device: Mini-FLOTAC
Device: Crypto/Giardia Duo Strip
Procedure: Formalin-ether concentration technique
Device: CCA RDT
Procedure: Koga agar plate culture
Procedure: Kinyoun staining
Device: Multiplex PCR
Procedure: Metagenomics analysis

SUMMARY:
NIDIAG is an international collaboration on integrated diagnosis-treatment platforms, funded by the European Commission (EC). NIDIAG aims to develop an improved, patient-centred system for delivering primary health care in resource-constrained settings. NIDIAG will investigate three clinical syndromes, namely (i) persistent digestive disorders, (ii) persistent fever and (iii) neurological disorders, due to neglected tropical diseases (NTDs). The current study focuses on persistent digestive disorders, which are defined as diarrhoea or abdominal pain that last for at least 2 weeks.

While acute diarrhoea has been studied globally, few research activities have focused on the epidemiology, diagnosis and treatment of long-lasting diarrhoeal episodes (2 weeks and longer) in the tropics. The spectrum of possibly involved pathogens includes more than 30 bacterial, parasitic and viral infectious agents. This lack of data may be explained by the fact that people suffering from NTDs might only seek care at a late stage of the disease. Furthermore, health systems in affected regions are often weak and their primary health-care centres are often under-staffed and lack essential diagnostic equipment.

The hypothesis of this study is that development of an evidence-based syndromic approach can lead to better diagnosis and management of NTDs in patients with persistent digestive disorders. The study will be carried out in two West African countries (Côte d'Ivoire and Mali) and in two Asian countries (Indonesia and Nepal). The study will follow a "case-control" design and patients and controls will be prospectively enrolled. In order to address the knowledge gaps, three specific objectives will be pursued. First, the contribution of NTDs to the 'persistent digestive disorders syndrome' will be assessed. Second, the value of clinical features and rapid diagnostic tests (RDTs) for the diagnosis of target NTDs that give rise to persistent digestive disorders will be determined. Third, the clinical response to standard empiric and targeted treatment of several NTDs in patients with persistent digestive disorders will be evaluated. These objectives will provide a long-term benefit for the communities by improving the clinical decision-making process for the target NTDs and thus, better diagnostic work-up and patient management can be achieved in the study countries and other similar resource-constrained countries

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged ≥1 year presenting with persistent diarrhoea (≥3 loose stools per days for ≥2 weeks; symptomatic group) and/or children (aged 1-18 years) with persistent abdominal pain (localized or diffuse abdominal pain lasting for ≥2 weeks, with possible intermittence/recurrence).
2. Individuals with written informed consent provided.

Exclusion Criteria:

1. Individuals in need of immediate intensive or surgical care.
2. Individuals who are unable or unwilling to give written informed consent.
3. Individuals who do not meet the inclusion criteria for being a case or control (e.g. people with acute diarrhoea).
4. Individuals with clinical jaundice (assessed by direct observation of the conjunctivae).
5. Individuals who are unable, in the study physician's opinion, to comply with the study requirements.
6. Individuals who are already participating in other ongoing diagnostic studies and/or clinical trials.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals aged ≥1 year presenting with persistent diarrhoea (≥3 loose stools per days for ≥2 weeks; symptomatic group) and/or children (aged 1-18 years) with persistent abdominal pain (localized or diffuse abdominal pain lasting for ≥2 weeks, with possible intermittence/recurrence) will be recruited together with matched controls.
Sampling Method: Probability Sample
Enrollment: 2800 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of neglected tropical diseases (NTDs) causing persistent digestive disorders (≥2 weeks) | 18 months
  The frequency, distribution, and if possible, intensity of target NTDs

SECONDARY OUTCOMES:
Sensitivity, specificity, crude and adjusted likelihood ratios (LR) and predictive values (post-test probabilities) of clinical features and laboratory tests for the diagnosis of target NTDs | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jürg Utzinger, PhD, Principal Investigator — Swiss Tropical & Public Health Institute; Katja Polman, PhD, Principal Investigator — Institute of Tropical Medicine, Belgium; Marleen Boelaert, PhD, Study Director — Institute of Tropical Medicine, Belgium
Locations (7):
- Hôpital Méthodiste de Dabou, Dabou, Côte d’Ivoire
- Indonesia (2):
  - Tulehu health center, Maluku Tengah, Maluku
  - Tulehu hospital, Maluku Tengah, Maluku
- Mali (2):
  - Institut National de Recherche en Santé Publique, Bamako
  - Niono District Reference Health Centre, Niono
- Nepal (2):
  - Dhankuta District Hospital, Dhankutā
  - B.P. Koirala Institute of Health Sciences, Dharān

REFERENCES:
- [Derived] Kristanti H, Meyanti F, Wijayanti MA, Mahendradhata Y, Polman K, Chappuis F, Utzinger J, Becker SL, Murhandarwati EEH. Diagnostic comparison of Baermann funnel, Koga agar plate culture and polymerase chain reaction for detection of human Strongyloides stercoralis infection in Maluku, Indonesia. Parasitol Res. 2018 Oct;117(10):3229-3235. doi: 10.1007/s00436-018-6021-5. Epub 2018 Aug 3. PMID 30074085
- [Derived] Polman K, Becker SL, Alirol E, Bhatta NK, Bhattarai NR, Bottieau E, Bratschi MW, Burza S, Coulibaly JT, Doumbia MN, Horie NS, Jacobs J, Khanal B, Landoure A, Mahendradhata Y, Meheus F, Mertens P, Meyanti F, Murhandarwati EH, N'Goran EK, Peeling RW, Ravinetto R, Rijal S, Sacko M, Saye R, Schneeberger PH, Schurmans C, Silue KD, Thobari JA, Traore MS, van Lieshout L, van Loen H, Verdonck K, von Muller L, Yansouni CP, Yao JA, Yao PK, Yap P, Boelaert M, Chappuis F, Utzinger J. Diagnosis of neglected tropical diseases among patients with persistent digestive disorders (diarrhoea and/or abdominal pain >/=14 days): Pierrea multi-country, prospective, non-experimental case-control study. BMC Infect Dis. 2015 Aug 18;15:338. doi: 10.1186/s12879-015-1074-x. PMID 26282537
- See also: A pre-study for this trial — http://www.controlled-trials.com/ISRCTN86951400/